CLINICAL TRIAL: NCT03829267
Title: eFIT: An Internet-based Intervention to Increase Physical Activity in Persons With Multiple Sclerosis
Brief Title: eFIT: An Internet-based Intervention to Increase Physical Activity in Persons With MS
Acronym: eFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Victoria M. Leavitt, Assistant Professor of Neuropsychology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAR4052-2
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Multiple Sclerosis
Keywords: exercise; physical activity
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to (a) SNAP treatment, (b) active control condition (eJournaling), or (c) waitlist control
Who Masked: Investigator
Masking Description: Participants will be enrolled in an internet-based intervention to increase physical activity. Only the PI will know whether participants are in the SNAP or eJournal condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eFIT Behavioral Intervention (Experimental): Intervention: Participants randomized to the eFIT condition will join a 1-hour peer group meeting online each week, called eFIT intervention. They will learn about accountability partners, and use the group as an accountability partner to state and attain physical fitness goals.
  Interventions: Behavioral: eFIT Intervention; Behavioral: Treatment as usual
- eJournal Behavioral Intervention (Active Comparator): Intervention: Participants in the eJournal condition will spend 1-hour online each week engaged in an active journaling activity, called eJournal Intervention. They will also receive the same psychoeducational materials online as the eFIT participants are presented in group.
  Interventions: Behavioral: eJournal Intervention; Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: eFIT Intervention — eFIT: social network accountability partners, a psychosocial intervention to increase physical activity in persons with multiple sclerosis
  Arms: eFIT Behavioral Intervention
Behavioral: eJournal Intervention — 1-hour online each week engaged in an active journaling activity
  Arms: eJournal Behavioral Intervention
Behavioral: Treatment as usual — Participants in this condition will complete baseline and follow-up surveys with the same frequency as the active treatment groups, but will receive neither eFIT nor eJournal.

SUMMARY:
eFIT is a technology-enabled internet based psychosocial intervention to increase physical activity in persons with multiple sclerosis, who are at unique risk for sedentary behaviors and for whom exercise and physical activity hold many benefits.

DETAILED DESCRIPTION:
This is a randomized controlled trial of an internet-based intervention to increase physical activity in persons with multiple sclerosis. Multiple sclerosis (MS) is the most common non-traumatic neurological cause of disability in young adults. Sedentary behavior, now recognized as a major contributor to increased morbidity is seen at higher rates and related to adverse health outcomes for persons with MS (PwMS). Prominent symptoms of MS (motor impairment, fatigue, depressed mood, pain), place this population at unique risk for increased sedentary behavior. And importantly, with increased age comes increased risk: patients over 60 are significantly more sedentary than middle-aged patients. On a positive note, current disease modifying therapies prolong time to disease progression, widening the window of opportunity for implementing behavioral interventions that support health and successful aging. Behaviors adopted early in life are more likely to be maintained into later adulthood. Physical activity is beneficial for PwMS on multiple levels: improved gait and balance, improved cognition, reduced depression and fatigue. Finding ways to increase physical activity is a key research priority for MS. Behavioral change is difficult to adopt and even more difficult to maintain. Here, we introduce a novel behavioral intervention to increase physical activity, eFIT, a technology-enabled (i.e., internet-delivered) support group-based treatment that leverages accountability to motivate and sustain behavioral change. Accountability constitutes the bedrock underlying the single most pervasive, successful, and widely embraced behavioral intervention known: Alcoholics Anonymous (AA). Through sponsors and support groups, AA utilizes accountability partners to deliver, reinforce, and sustain life-saving behavioral change. Here, we leverage accountability partners to motivate enduring behavioral change in physical activity participation, one of the single most difficult health behaviors to implement and maintain.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Diagnosis of multiple sclerosis

Exclusion Criteria:

* Cannot be available for the next 12 weeks consecutively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2020-04-13 (Actual); Study Completion 2020-04-13 (Actual)

PRIMARY OUTCOMES:
Adherence rate: Percentage of weekly eFIT group meetings that participants attend | 12-weeks
  Assess feasibility of the program: Acceptability of intervention based on attendance rates of participants meeting the criteria of attendance at two-thirds of the meetings over 12-weeks
Completion rate: Percentage of enrolled participants who complete follow-up questionnaires | 12-weeks
  Assess feasibility of the program: to retain and obtain completed questionnaires at immediate follow-up from two-thirds of enrolled participants meeting the criteria of two-thirds attendance.

SECONDARY OUTCOMES:
Change in International Physical Activity Questionnaire (IPAQ) total score (self-reported physical activity level) | 12-weeks
  International Physical Activity Questionnaire (IPAQ)-Long form includes 27 items divided into 5 subscales. For this trial, the total minutes/hours/days for items 1-25 will be calculated. Higher scores indicate more time spent engaged in physical activity. Items 26 and 27 will be excluded in the variable because they query about time spent sitting.
Patient Health Questionnaire-9 (PHQ-9) | 12-weeks
  Assess efficacy of the program to improve mood as defined by an increase in total score on PHQ-9. The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. Total score ranges from 0 to 27, with higher scores indicating worse depression.
UCLA Loneliness Scale | 12-weeks
  Assess efficacy of the program to decrease loneliness as defined by a decrease in total score on UCLA Loneliness Scale. This name never appears as anything other than UCLA Loneliness Scale, i.e. Russell 1996). Total score ranges from 0 to 60, with higher scores indicating worse loneliness.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Leavitt, MD, Principal Investigator — Assistant Professor of Neuropsychology
Locations (1):
- Columbia University Multiple Sclerosis Clinical Care and Research, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pate RR, Pratt M, Blair SN, Haskell WL, Macera CA, Bouchard C, Buchner D, Ettinger W, Heath GW, King AC, et al. Physical activity and public health. A recommendation from the Centers for Disease Control and Prevention and the American College of Sports Medicine. JAMA. 1995 Feb 1;273(5):402-7. doi: 10.1001/jama.273.5.402. PMID 7823386
- [Derived] Leavitt VM, Aguerre IM, Lee N, Riley CS, De Jager PL, Bloom S. RCT of a Telehealth Group-Based Intervention to Increase Physical Activity in Multiple Sclerosis: eFIT. Neurol Clin Pract. 2021 Aug;11(4):291-297. doi: 10.1212/CPJ.0000000000001039. PMID 34484928